CLINICAL TRIAL: NCT00348725
Title: An Open Label, Parallel-Arm, Multicenter Trial Assessing the Acceptability of 4 Dosages of a New Fixed Dose Combination of Fenofibrate and Metformin in Patients With Type 2 Diabetes and Dyslipidemia
Brief Title: Acceptability of a Fixed Combination of Fenofibrate and Metformin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C LF23-0121 04 02
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2007-09-03 (Estimated); Status verified 2007-08

CONDITIONS: Dyslipidemia/Glucose Metabolism Disorder
Keywords: Treatment of Dyslipidemia and of Type 2 Diabetes Mellitus
MeSH Terms: conditions — Dyslipidemias; Glucose Metabolism Disorders | interventions — Fenofibrate; Pharmaceutical Preparations

INTERVENTIONS:
Drug: fenofibrate and metformin fixed combination (drug)

SUMMARY:
The primary objective was to assess the acceptability of a 4-week treatment of 4 new fixed-dose combinations of fenofibrate and metformin, in patients with type 2 diabetes and dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus and dyslipidemia.

Exclusion Criteria:

* Type 1 diabetes, uncontrolled type 2 diabetes, - HbA1c ≥ 10 % - Fasting plasma glucose > 300 mg/dL - Triglycerides > 500 mg/dL

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69
Dates: Start 2005-04

PRIMARY OUTCOMES:
Quotation by Visual Numeric Rating Scale before and after 4-week treatment

SECONDARY OUTCOMES:
Assessment of safety by reporting of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (25):
- France (25):
  - Site 24, Anzin
  - Site 23, Bachant
  - Site 21, Bauné
  - Site 32, Bersée
  - Site 34, Briollay
  - Site 27, Denain
  - Site 28, Denain
  - Site 5, Le Temple-de-Bretagne
  - Site 29, Nantes
  - Site 2, Nantes
  - Site 8, Nantes
  - Site 9, Nantes
  - Site 1, Nort-sur-Erdre
  - Site 13, Parçay-les-Pins
  - Site 26, Quarouble
  - Site 7, Saint Aignan Le Grand
  - Site 30, Saint-Amand
  - Site 10, Saint-Étienne-de-Montluc
  - Site 4, Saint-Herblain
  - Site 11, Sautron
  - Site 17, Segré
  - Site 33, Thiant
  - Site 12, Thouars
  - Site 25, Vieux-Condé
  - Site 20, Vihiers